CLINICAL TRIAL: NCT05949775
Title: Clinical Study on the Treatment of Advanced Malignant Solid Tumors With the Combination of mRNA
Brief Title: Clinical Study of mRNA Vaccine in Patients With Advanced Malignant Solid Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stemirna Therapeutics (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-06-mRNA-COM
Record Dates: First submitted 2023-06-28; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Advanced Malignant Solid Tumors

STUDY DESIGN:
Intervention Model Description: PD-1/PD-L1 drug therapy benefits patients with secondary drug-resistant malignant solid tumors, including but not limited to gastric cancer, esophageal cancer, and other gastrointestinal tumors of MSI-H.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Neoantigen mRNA Personalised Cancer in combination with Stintilimab Injection. Participants will receive a total of 9 cycles of PCV every 21 days
  Interventions: Biological: Neoantigen mRNA Personalised Cancer vaccine

INTERVENTIONS:
Biological: Neoantigen mRNA Personalised Cancer vaccine — Drug: Neoantigen mRNA Personalised Cancer vaccine in combination with Stintilimab Injection Subcutaneous Injection

SUMMARY:
This study is an open, single arm, dose increasing study to evaluate the safety and efficacy of the combination of mRNA personalized tumor vaccine encoding neoantigen (hereinafter referred to as tumor vaccine) and Sintilimab injection (hereinafter referred to as Sintilimab) in the treatment of advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥18 years old, without limitation of sex at time of consent.
* Patients with malignant solid tumors confirmed by histopathology or cytology and having at least one measurable lesion.
* Fresh biopsy specimens can be provided for vaccine preparation.
* Patients with malignant solid tumors who develop secondary drug resistance after receiving PD-1/PD-L1 drug therapy, including but not limited to gastric cancer, esophageal cancer, and other gastrointestinal tumors of MSI-H

Exclusion Criteria:

* It is known that it is allergic to any tumor vaccine and Sintilimab preparations; Or have experienced severe allergic reactions to other monoclonal antibodies in the past;
* The predicted number of new antigens is less than 10;
* Those who are pregnant or breastfeeding;
* Those with an expected survival period of less than 3 months;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | Time Frame: from enrolling to patients disease progression，assessed up to 24 months